CLINICAL TRIAL: NCT01079026
Title: Functional Outcome After Lumbar Epidural Steroid Injection
Brief Title: Outcome After Lumbar Epidural Steroid Injection
Status: Completed | Type: Observational
Sponsor: Scuderi, Gaetano J., M.D. (Other)
Collaborators: Cytonics Corporation (Industry)
Responsible Party: Gaetano J Scuderi, MD, Stanford University
Other Study IDs: CYt.003
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Disc Disease
Keywords: biomarker; epidural steroid; radiculopathy; hnp
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lavage fluid from epidural space
Oversight: Data Monitoring Committee: Yes

SUMMARY:
prospectively validate a fibronectin-aggrecan complex as a biomarker for response to ESI for radiculopathy with HNP

DETAILED DESCRIPTION:
We will measure levels of the protein complex in the epidural space of patients undergoing lumbar ESI for radiculopathy with HNP. We assess functional outcomes at baseline and after treatment with the Medical Outcomes Study Short Form-36 instrument (SF-36). Our hypothesis was that the complex is present in patients with clinically significant functional improvement after ESI.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of sensory symptoms with the primary complaint as pain as well as varying sensory symptoms (e.g. tingling, numbness) in one or more lumbar nerve root distributions
* Positive physical exam findings including sensory findings consistent with a spinal nerve root, a positive straight leg raise test, and/or a diminished patellar or Achilles DTR consistent with sensory symptoms; AND
* MRI of lumbar spine positive for HNP in a distribution correlating with physical examination

Exclusion Criteria:

* Plain radiography demonstrating severe loss of disc height, high grade DDD, spondylolisthesis greater than grade I
* A history of prior lumbar surgery or trauma, weakness in a consistent distribution (non-progressive with strength at least 4/5)
* Red flags including progressive weakness, bowel/bladder complaints, radiographic unknown mass, unexpected weight loss; AND
* Diagnosis of inflammatory arthritides, crystalline arthropathies, or other rheumatologic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered candidates for ESI were 18 years of age or greater with a history of leg sensory complaints primarily dictated by pain with associated sensory symptoms and/or low back pain for two weeks or more who had failed expectant management with NSAIDS, activity modification, and/or physical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
functional outcome on SF-36 following ESI | 2-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano J Scuderi, MD, Principal Investigator — Stanford University